CLINICAL TRIAL: NCT00401362
Title: A Double-Blind Placebo-Controlled Study of Methylnaltrexone (MNTX) for the Relief of Constipation Due to Chronic Opioid Therapy in Patients With Advanced Medical Illness
Brief Title: A a Single Dose Efficacy Study in Inducing Laxation in Advance Illness Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Tage Ramakrishna, MD, Progenics Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MNTX 301
Record Dates: First submitted 2006-11-16; First posted 2006-11-20 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Advanced Illness Patients With Opioid Induced Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: SC Methylnaltrexone
- Arm 3 (Placebo Comparator)
  Interventions: Drug: SC Placebo
- Arm 2 (Experimental)
  Interventions: Drug: SC Methylnaltrexone

INTERVENTIONS:
Drug: SC Methylnaltrexone — Dose 1
  Arms: Arm 1
Drug: SC Placebo
  Arms: Arm 3
Drug: SC Methylnaltrexone — Dose 2
  Arms: Arm 2

SUMMARY:
To test the effectiveness of MNTX in advanced illness subjects.

DETAILED DESCRIPTION:
To determine the efficacy of MNTX compared to placebo to induce laxation in patients receiving opioids.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced medical illness with a life expectancy of 1 to 6 months
2. No clinically significant laxation within 48 hours prior to the first dose of study drug
3. On stable opioid and laxative regimen for a least 3 days prior to treatment
4. Age greater than 18years
5. Females of child-bearing age must have a negative pregnancy test.

Exclusion Criteria:

1. Females who are pregnant or nursing.
2. Previous treatment with MNTX or prior treatment with naltrexone or naloxone for treatment of OIC
3. Any disease process suggestive of gastrointestinal obstruction
4. Fecal ostomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2003-02; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Efficacy of SC MNTX compared with placebo in inducing laxation | 29 days
  The primary objective is to determine the efficacy of SC MNTX administered as a single dose, dose 1 and dose 2 compared with placebo in inducing laxation in 4 hours in patients with advanced medical illness and OIC who are poorly responsive to laxatives.

CONTACTS AND LOCATIONS:
Overall Officials: Tage Ramakrishna, MD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (1):
- Progenics Pharmaceuticals, Inc., Tarrytown, New York, United States

REFERENCES:
- [Derived] Chamberlain BH, Rhiner M, Slatkin NE, Stambler N, Israel RJ. Subcutaneous methylnaltrexone for opioid-induced constipation in advanced-illness patients with or without active cancer. Pain Manag. 2020 Mar;10(2):73-84. doi: 10.2217/pmt-2019-0045. Epub 2020 Jan 17. PMID 31951150
- [Derived] Janku F, Johnson LK, Karp DD, Atkins JT, Singleton PA, Moss J. Treatment with methylnaltrexone is associated with increased survival in patients with advanced cancer. Ann Oncol. 2016 Nov;27(11):2032-2038. doi: 10.1093/annonc/mdw317. Epub 2016 Aug 29. PMID 27573565
- [Derived] Nalamachu SR, Pergolizzi J, Taylor R Jr, Slatkin NE, Barrett AC, Yu J, Bortey E, Paterson C, Forbes WP. Efficacy and Tolerability of Subcutaneous Methylnaltrexone in Patients with Advanced Illness and Opioid-Induced Constipation: A Responder Analysis of 2 Randomized, Placebo-Controlled Trials. Pain Pract. 2015 Jul;15(6):564-71. doi: 10.1111/papr.12218. Epub 2014 May 10. PMID 24815199
- [Derived] Slatkin N, Thomas J, Lipman AG, Wilson G, Boatwright ML, Wellman C, Zhukovsky DS, Stephenson R, Portenoy R, Stambler N, Israel R. Methylnaltrexone for treatment of opioid-induced constipation in advanced illness patients. J Support Oncol. 2009 Jan-Feb;7(1):39-46. PMID 19278178